CLINICAL TRIAL: NCT05607238
Title: Patient Perspective of Midline Catheters Versus Ultrasound Guided Peripheral IVs for Difficult IV Access in the ED
Brief Title: Patient Perspective Midline Catheter in the Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the key physicians is leaving the institution and other delays have put us behind our timeline. We do not intend to proceed with the trial at this time.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00089914
Record Dates: First submitted 2022-10-13; First posted 2022-11-07 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-10

CONDITIONS: Patient Satisfaction; Patient Preference
Keywords: IV access; ultrasound guided IV; emergency care
MeSH Terms: conditions — Patient Satisfaction; Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Peripheral IV (Active Comparator): Placement of 4-5cm angiocath under ultrasound guidance
  Interventions: Procedure: Ultrasound Guided Vascular Access - peripheral IV
- Ultrasound Guided Midline Catheter (Experimental): Placement of 10-15cm midline catheter under ultrasound guidance
  Interventions: Procedure: Ultrasound Guided Vascular Access - Midline catheter

INTERVENTIONS:
Procedure: Ultrasound Guided Vascular Access - Midline catheter — Ultrasound guided vascular access with a midline IV catheter
  Arms: Ultrasound Guided Midline Catheter
Procedure: Ultrasound Guided Vascular Access - peripheral IV — Ultrasound guided vascular access with a peripheral IV catheter
  Arms: Ultrasound Guided Peripheral IV

SUMMARY:
This study examines the patient satisfaction and perspective on the use of ultrasound guided midline intravenous catheters compared to standard ultrasound guided peripheral catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the emergency department
* Failed 2 or more conventional attempts at vascular access *or*
* history of requiring US guided vascular access
* US Fellowship trained physician available

Exclusion Criteria:

* basilic vein access is contraindicated
* patient undergoing advanced resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction with Procedure | Immediately after procedure/Baseline
  Score describes a patient's satisfaction with a healthcare decision. It measures satisfaction across 6 domains via 6 questions scored on a 5 point scale. Score ranges from 6 to 30. A low score signifies dissatisfaction, a high score signifies high satisfaction.
Patient Satisfaction with Procedure | At 48 Hours Post Baseline
  Score describes a patient's satisfaction with a healthcare decision. It measures satisfaction across 6 domains via 6 questions scored on a 5 point scale. Score ranges from 6 to 30. A low score signifies dissatisfaction, a high score signifies high satisfaction.

SECONDARY OUTCOMES:
Number of needle punctures in a 24 hour period (patient reported) | up to 48 hours
Duration of Successful Access | up to 48 hours
  IV/Cath dwell time in hours
Number of Needle Sticks | up to 48 hours
  Prior to gaining successful access
Number of Insertion Attempts | up to 48 hours
  For ultrasound guided access
Emergency Department (ED) Length of Stay | up to 48 hours
  in hours
Hospital Length of Stay | up to 48 hours
  in hours
Patient Satisfaction | immediately post intervention/baseline and at 48 hours past baseline
  this is a single question measuring satisfaction with the intervention overall on a Likert Scale 1-10,
Number of Insertion Related Complications | up to 48 hours
  Includes failed attempts, arterial punctures, infiltrations, hematoma formations
Number of Dwell Related Complications | up to 48 hours
  Includes inability to flush, catheter dislodgement, leakage around the catheter site, insertion site erythema, insertion site pain, drainage from catheter, edema, ecchymosis, superficial thrombosis, Deep vein thrombosis (DVT), line associated infection, vesicant extravasation, skin necrosis, neurovascular injury, arterial injury
Time to Access | up to 24 hours
  minutes from procedure start to procedure completion

CONTACTS AND LOCATIONS:
Overall Officials: Casey Glass, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No